CLINICAL TRIAL: NCT06102005
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose Ranging Study to Assess the Efficacy, Safety, and Tolerability of Subcutaneous Lunsekimig in Adult Participants With Moderate-to-severe Asthma
Brief Title: Dose Ranging Study of Lunsekimig Compared With Placebo-control in Adult Participants With Moderate-to-severe Asthma
Acronym: AIRCULES
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRI16762; U1111-1280-5514 (Other: WHO); 2023-503712-33 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Lunsekimig Dose1 interval 1 (Experimental): Participants will receive Dose 1 of lunsekimig (subcutaneous injection) according to established dosing interval 1
  Interventions: Drug: Lunsekimig
- Lunsekimig Dose 1 interval 2 (Experimental): Participants will receive Dose 1 of lunsekimig (subcutaneous injection) according to established dosing interval 2
  Interventions: Drug: Lunsekimig
- Lunsekimig Dose 2 interval 1 (Experimental): Participants will receive Dose 2 of lunsekimig (subcutaneous injection) according to established dosing interval 1
  Interventions: Drug: Lunsekimig
- Lunsekimig Dose 2 interval 2 (Experimental): Participants will receive Dose 2 of lunsekimig (subcutaneous injection) according to established dosing interval 2
  Interventions: Drug: Lunsekimig
- Placebo (Placebo Comparator): Participants will receive placebo (subcutaneous injection) according to established dosing intervals corresponding to Dose 1 and Dose 2
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lunsekimig — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: Lunsekimig Dose 1 interval 2; Lunsekimig Dose 2 interval 1; Lunsekimig Dose 2 interval 2; Lunsekimig Dose1 interval 1
Drug: Placebo — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: Placebo

SUMMARY:
This is a Phase 2b, global, multicenter, randomized, double-blind, placebo-controlled, parallel group, dose ranging study to assess the efficacy, safety, and tolerability of add-on therapy with SC lunsekimig in adult participants aged 18 to 80 years, (inclusive) with moderate-to-severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* A physician-diagnosed moderate-to-severe asthma for ≥12 months based on GINA guidelines Steps 4 and 5
* Participants with existing treatment with moderate-to-high doses of ICS therapy for in combination with at least 1 but no more than 2 additional controller medications at least 3 months with a stable dose ≥1 month prior to Visit 1
* At least 1 asthma exacerbation in the past year, with at least one exacerbation occurring while on treatment with moderate to high doses of ICS therapy
* ACQ-5 score more than 1.5 at Screening (Visit 1)

Exclusion Criteria:

* Chronic obstructive or other lung diseases (eg, COPD, idiopathic pulmonary fibrosis, etc) which may impair lung function, or another diagnosed pulmonary or systemic disease.
* Current smoker or former smoker with cessation within 6 months of Screening or history of >10 pack-years. Active vaping of any products and/or marijuana smoking within 6 months of Screening.
* Participants who experience a deterioration of asthma that results in emergency treatment or hospitalization, or treatment with systemic steroids within 1 month prior to the Screening
* Participants who have experienced an upper or lower respiratory tract infection within the 4 weeks prior to Screening
* For participants on chronic OCS use for the maintenance treatment of asthma: history of a serious infection requiring hospitalization within the past 12 months prior to Randomization (Visit 2).
* Participants with active tuberculosis (TB), latent TB, a history of incompletely treated TB, suspected extrapulmonary TB infection, or who are at high risk of contracting TB (such as close contact with individuals with active or latent TB) or received Bacillus Calmette-Guérin (BCG)-vaccination within 12 weeks prior to Screening
* Severe concomitant illness that would in the Investigator's opinion inhibit the participant's participation in the study, including for example, but not limited to, hypertension, renal disease, neurological conditions, heart failure and pulmonary disease
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of asthma exacerbation events | From baseline to week 48

SECONDARY OUTCOMES:
Change from baseline in pre-bronchodilator (BD) FEV1 | From baseline to week 48
Change from baseline in post-BD FEV1 | From baseline to week 48
The absolute change in the percent predicted FEV1 from baseline (pre-BD and post-BD) | From baseline to week 48
Proportion of participants with ≥ 0.5-point reduction in ACQ-5 score | From baseline to week 48
  ACQ-5 is Asthma control questionnaire assessing symptoms. Lower score shows better asthma control
Change from baseline in ACQ-5 score | From baseline to week 48
Change from baseline in FeNO | From baseline to week 48
Time to first asthma exacerbation | From baseline to week 48
Annualized rate of severe asthma exacerbations requiring hospitalization or emergency room or urgent care visit | From baseline to week 48
Average number of inhalations per day of short-acting beta 2-agoinst (SABA), Low dose ICS/formoterol or ICS/SABA for symptom relief | From baseline to week 48
Change from baseline in St. George's Respiratory Questionnaire (SGRQ) scores | From baseline to week 48
  Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating more limitations.
Proportion of participants with ≥4-point improvement in SGRQ score | From baseline to week 48
Change from baseline in Asthma Quality of Life Questionnaire Standardized for 12 years and older (AQLQ{S} +12) scores | From baseline to week 48
Proportion of participants with ≥0.5-point improvement in AQLQ(S)+12 domain and total scores | From baseline to week 48
Change from baseline in ACQ scores | From baseline to week 48
Proportion of participants with ≥0.5-point reduction in ACQ-6 and ACQ-7 score | From baseline to week 48
Serum lunsekimig concentrations | From baseline to week 52
Anti-drug antibodies (ADA) against lunsekimig | From baseline to week 52
Incidence of participants with treatment-emergent adverse events (TEAEs), including local reactions, adverse events of special interests (AESIs), serious adverse events (SAEs) | From baseline to week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinial Science & Operations, Study Director — Sanofi
Locations (156):
- United States (48):
  - Allergy, Asthma & Immunology Associates- Site Number : 8400009, Scottsdale, Arizona
  - Yuma Pulmonary & Sleep Research, LLC- Site Number : 8400072, Yuma, Arizona
  - Antelope Valley Clinical Trials- Site Number : 8400020, Lancaster, California
  - Amicis Research Center - Northridge - Nordhoff Street- Site Number : 8400032, Northridge, California
  - Optimus Medical- Site Number : 8400046, San Francisco, California
  - Allergy and Asthma Associates of Santa Clara Valley Research Center- Site Number : 8400038, San Jose, California
  - Clinical Trials Management Services - Thousand Oaks- Site Number : 8400053, Thousand Oaks, California
  - Allianz Research Institute CO- Site Number : 8400026, Aurora, Colorado
  - Velocity Clinical Research - Denver- Site Number : 8400027, Englewood, Colorado
  - Western States Clinical Research- Site Number : 8400014, Wheat Ridge, Colorado
  - Beautiful Minds Clinical Research Center- Site Number : 8400049, Cutler Bay, Florida
  - Qway Research - Hialeah- Site Number : 8400015, Hialeah, Florida
  - Clintex Research Group - Miami - Coral Way- Site Number : 8400048, Miami, Florida
  - High Quality Research- Site Number : 8400039, Miami, Florida
  - Innovations Biotech- Site Number : 8400040, Miami, Florida
  - New Access Medical Center- Site Number : 8400043, Miami, Florida
  - Deluxe Health Center- Site Number : 8400045, Miami Lakes, Florida
  - Advanced Research Institute - New Port Richey- Site Number : 8400044, New Port Richey, Florida
  - Pines Care Research Center- Site Number : 8400057, Pembroke Pines, Florida
  - Windom Allergy, Asthma and Sinus Specialists- Site Number : 8400019, Sarasota, Florida
  - Appalachian Clinical Research- Site Number : 8400050, Calhoun, Georgia
  - PMG Research of Christie Clinic- Site Number : 8400066, Champaign, Illinois
  - Velocity Clinical Research Lafayette Site Number : 8400060, Lafayette, Louisiana
  - Javara - Privia Medical Group - Annapolis- Site Number : 8400033, Annapolis, Maryland
  - Brigham & Women's Hospital- Site Number : 8400034, Boston, Massachusetts
  - University of Michigan Health System - Ann Arbor- Site Number : 8400004, Ann Arbor, Michigan
  - Javara - Mankato Clinic- Site Number : 8400051, Mankato, Minnesota
  - Midwest Clinical Research Center - St. Louis- Site Number : 8400006, St Louis, Missouri
  - Circuit Clinical - Middletown Medical - 111 Maltese Drive- Site Number : 8400065, Middletown, New York
  - Icahn School of Medicine at Mount Sinai- Site Number : 8400058, New York, New York
  - Carolina Clinical Research - Charlotte- Site Number : 8400071, Charlotte, North Carolina
  - Tryon Medical Partners - Charlotte - Piedmont Row Drive South- Site Number : 8400029, Charlotte, North Carolina
  - Clinical Research Of Gastonia- Site Number : 8400013, Gastonia, North Carolina
  - Bernstein Clinical Research Center- Site Number : 8400016, Cincinnati, Ohio
  - Asthma & Allergy Center - Toledo- Site Number : 8400017, Toledo, Ohio
  - OK Clinical Research- Site Number : 8400021, Edmond, Oklahoma
  - Velocity Clinical Research - Medford- Site Number : 8400059, Medford, Oregon
  - Clinical Research Associates of Central PA - Dubois- Site Number : 8400069, DuBois, Pennsylvania
  - Allergy & Clinical Immunology Associates Pittsburgh- Site Number : 8400007, Pittsburgh, Pennsylvania
  - Circuit Clinical - PMSI Comprehensive Healthcare for Life - Pottstown - Medical Drive- Site Number : 8400064, Pottstown, Pennsylvania
  - VitaLink Research - Anderson - East Greenville- Site Number : 8400063, Anderson, South Carolina
  - Velocity Clinical Research - Charleston- Site Number : 8400061, Charleston, South Carolina
  - Orion Clinical Research- Site Number : 8400001, Austin, Texas
  - South Texas Medical Research Institute - TTS Research- Site Number : 8400010, Boerne, Texas
  - Baylor University Medical Center- Site Number : 8400002, Dallas, Texas
  - Western Sky Medical Research- Site Number : 8400023, El Paso, Texas
  - Metroplex Pulmonary and Sleep Center- Site Number : 8400022, McKinney, Texas
  - VAST Clinical Research- Site Number : 8400062, Plano, Texas
- Argentina (10):
  - Investigational Site Number : 0320007, Berazategui, Buenos Aires
  - Investigational Site Number : 0320003, La Plata, Buenos Aires
  - Investigational Site Number : 0320002, Rosario, Santa Fe Province
  - Investigational Site Number : 0320006, Rosario, Santa Fe Province
  - Investigational Site Number : 0320005, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320009, Mendoza
  - Investigational Site Number : 0320008, San Miguel de Tucumán
  - Investigational Site Number : 0320010, Santa Fe
- Brazil (8):
  - Associacao Proar- Site Number : 0760003, Salvador, Estado de Bahia
  - Universidade Federal de Goias- Site Number : 0760007, Goiânia, Goiás
  - Centro de Estudos em Terapias Inovadoras- Site Number : 0760002, Curitiba, Paraná
  - Inst de Medicina Integral Professor Fernando Figueira- Site Number : 0760009, Recife, Pernambuco
  - Hospital São Lucas da PUCRS - Porto Alegre - Avenida Ipiranga- Site Number : 0760001, Porto Alegre, Rio Grande do Sul
  - Hospital Dia do Pulmão- Site Number : 0760005, Blumenau, Santa Catarina
  - CCBR / IBPClin - Instituto Brasil de Pesquisa Clínica- Site Number : 0760006, Rio de Janeiro
  - Incor - Instituto do Coracao- Site Number : 0760011, São Paulo
- Canada (4):
  - Investigational Site Number : 1240003, Hamilton, Ontario
  - Investigational Site Number : 1240005, Stoney Creek, Ontario
  - Investigational Site Number : 1240004, Sherbrooke, Quebec
  - Investigational Site Number : 1240001, Trois-Rivières, Quebec
- Chile (9):
  - Investigational Site Number : 1520010, Valdivia, Los Ríos Region
  - Investigational Site Number : 1520001, Talca, Maule Region
  - Investigational Site Number : 1520006, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520009, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520008, Quillota, Región de Valparaíso
  - Investigational Site Number : 1520011, Viña del Mar, Región de Valparaíso
- China (18):
  - Investigational Site Number : 1560011, Beijing
  - Investigational Site Number : 1560010, Changchun
  - Investigational Site Number : 1560017, Changsha
  - Investigational Site Number : 1560008, Chengdu
  - Investigational Site Number : 1560001, Guangzhou
  - Investigational Site Number : 1560009, Guangzhou
  - Investigational Site Number : 1560006, Hefei
  - Investigational Site Number : 1560014, Hohhot
  - Investigational Site Number : 1560018, Mianyang
  - Investigational Site Number : 1560007, Nanchang
  - Investigational Site Number : 1560002, Pingxiang
  - Investigational Site Number : 1560013, Shanghai
  - Investigational Site Number : 1560015, Shenyang
  - Investigational Site Number : 1560005, Wenzhou
  - Investigational Site Number : 1560003, Wuhan
  - Investigational Site Number : 1560004, Xuzhou
  - Investigational Site Number : 1560016, Yangzhou
  - Investigational Site Number : 1560012, Zhanjiang
- India (8):
  - Investigational Site Number : 3560002, Coimbatore
  - Investigational Site Number : 3560006, Delhi
  - Investigational Site Number : 3560009, Hyderabad
  - Investigational Site Number : 3560008, Kanpur
  - Investigational Site Number : 3560007, Kozhikode
  - Investigational Site Number : 3560003, Lucknow
  - Investigational Site Number : 3560001, Nagpur
  - Investigational Site Number : 3560004, Pune
- Israel (9):
  - Investigational Site Number : 3760006, Ashkelon
  - Investigational Site Number : 3760001, Haifa
  - Investigational Site Number : 3760008, Haifa
  - Investigational Site Number : 3760003, Jerusalem
  - Investigational Site Number : 3760002, Jerusalem
  - Investigational Site Number : 3760010, Petah Tikva
  - Investigational Site Number : 3760009, Ramat Gan
  - Investigational Site Number : 3760004, Rehovot
  - Investigational Site Number : 3760007, Tel Aviv
- Japan (10):
  - Investigational Site Number : 3920004, Kamogawa, Chiba
  - Investigational Site Number : 3920002, Sakaidechō, Kagawa-ken
  - Investigational Site Number : 3920010, Yokohama, Kanagawa
  - Investigational Site Number : 3920011, Chūō, Tokyo
  - Investigational Site Number : 3920005, Ube, Yamaguchi
  - Investigational Site Number : 3920008, Fukushima
  - Investigational Site Number : 3920003, Higashiōmi
  - Investigational Site Number : 3920006, Kyoto
  - Investigational Site Number : 3920009, Kyoto
  - Investigational Site Number : 3920012, Miyazaki
- Mexico (7):
  - Investigational Site Number : 4840001, Guadalajara, Jalisco
  - Investigational Site Number : 4840004, Monterrey, Nuevo León
  - Investigational Site Number : 4840005, San Juan del Río, Querétaro
  - Investigational Site Number : 4840002, Chihuahua City
  - Investigational Site Number : 4840003, Durango
  - Investigational Site Number : 4840007, Mérida
  - Investigational Site Number : 4840008, Veracruz
- South Africa (6):
  - Investigational Site Number : 7100004, Benoni
  - Investigational Site Number : 7100005, Benoni
  - Investigational Site Number : 7100003, Cape Town
  - Investigational Site Number : 7100002, Cape Town
  - Investigational Site Number : 7100001, Durban
  - Investigational Site Number : 7100006, Lochner ROAD
- South Korea (6):
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100005, Seoul
- Turkey (Türkiye) (7):
  - Investigational Site Number : 7920001, Akdeniz
  - Investigational Site Number : 7920006, Bursa
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920004, Izmir
  - Investigational Site Number : 7920005, İzmit
  - Investigational Site Number : 7920007, Kayseri
- United Kingdom (6):
  - Investigational Site Number : 8260001, Cambridge, Cambridgeshire
  - Investigational Site Number : 8260004, Glasgow, Edinburgh, City of
  - Investigational Site Number : 8260005, Chertsey, Surrey
  - Investigational Site Number : 8260003, Birmingham
  - Investigational Site Number : 8260008, Bradford
  - Investigational Site Number : 8260009, Bristol

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org